CLINICAL TRIAL: NCT05037578
Title: A Church-based Intervention for Increasing Screening for Dementia Among African American Older Adults (ADC Pilot): Project Grace
Brief Title: Encouraging Cognitive Screenings at African American Churches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2017382 KC
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Dementia; Healthy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Grace (Experimental): This intervention will be delivered through church-based multilevel activities by trained church leaders using religiously/ culturally-tailored study materials (sermon guides, responsive readings, educational games, brochures, educational/testimonial videos) packaged in a culturally-tailored. Intervention churches will receive the Project Grace Tool Kit and intervention implementation directions to seek cognitive screening. These churches will hold a Project Grace Kickoff event, where a sermon, and other tool kit materials will be distributed. After the Kick-off, liaisons will deliver 1-2 Tool Kit materials/activities per month through targeted multilevel church activities over 4 months. Delivery of intervention components will coincide with existing, multilevel activities that occur in churches through: a) church-wide services, b) outreach ministry groups; and c) individual level activities (e.g., text/voice/email health promotion messages from church) over 4 months.
  Interventions: Behavioral: Project Grace
- Standard Control (Active Comparator): Standard information churches will receive standard dementia education information. These churches will receive: a) non-tailored project materials collected from mental health organizations and b) standard community-based mental health screening events) coordinated by their Community Health Liaisons. These churches will receive all Project Grace Tool Kit materials and implementation training after the completion of assessments.
  Interventions: Behavioral: Project Grace

INTERVENTIONS:
Behavioral: Project Grace — A multilevel church-based intervention to encourage cognitive screens and brain health.

SUMMARY:
This pilot study plans to examine feasibility and outcomes of a culturally/religiously-tailored church-based dementia screening intervention among older adult African American church members and community members who use church outreach services in 4 African American churches.

DETAILED DESCRIPTION:
The primary aim of this study is to conduct an exploratory pilot study to examine feasibility and outcomes of a culturally/religiously-tailored church-based dementia screening intervention among older adult African American church members and community members who use church outreach services in 4 African American churches (N=100). Our secondary outcomes are to assess the impact of the intervention on dementia-related stigma and linkage to care. Intervention content is based on the Theory of Planned Behavior; intervention delivery is based on the Social-Ecological Model - both guided by a faith community engagement approach. Trained faith leaders will deliver the tailored intervention through multilevel church outlets: individual self-help resources (e.g., risk checklist, commitment to screening cards); group ministry discussion guides/seminar on dementia; church-wide services using sermon guides, responsive readings, and church bulletin inserts; and church-community level text messages, dementia screening, and linkage to care services. Two screening events will be held at each church. We will also conduct a process evaluation that will include post-test study focus groups.

Specific Aim 1. Test a religiously/culturally-tailored, church-based dementia screening intervention on receipt of dementia screening, stigma, and linkage to care use among an older adult African American church-populations at 4 months.

Hypothesis. The tailored church-based dementia screening intervention will evidence increased screening and linkage to care rates, and lower dementia-related stigma beliefs at 4 months.

Specific Aim 2. Evaluate predictors of receipt of dementia screening at 4 months among older adult African American church-populations to determine modifiable screening facilitators/barriers.

Specific Aim 3. Conduct a process evaluation to examine study intervention implementation facilitators, barriers, and dose along with exposure and satisfaction to identify essential intervention components.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55
2. Regular church member (attending church > monthly) or community member receiving church outreach services (>3 times annually)
3. Willing to participate in two surveys (baseline and 4 months)
4. Willing to provide contact information for at least 2 other persons
5. Residing in the Kansas City metropolitan area
6. Provide a working contact email address or number

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, UMKC, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Project Grace | Standard Control
Started | 62 | 37
Completed | 54 | 33
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project Grace | Standard Control | Total
Number analyzed (Participants) | 62 | 37 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.6) | 68.4 (8.3) | 68.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 31 | 82
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 60 | 35 | 95
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 37 | 99
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 37 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received a Cognitive Screening
Description: Question at 4 months from baseline asking whether the participant has received a cognitive screening within the last 4 months
Time Frame: 4 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Project Grace | Standard Control
Number analyzed (Participants) | 62 | 37
Participants | 5 | 11

2. Primary Outcome: Number of Participants Who Were Linked to Care Services
Description: Question at 4 months from baseline asking whether the participant has received a linkage to care services within the last 4 months
Time Frame: 4 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Project Grace | Standard Control
Number analyzed (Participants) | 62 | 37
Participants | 5 | 11

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Project Grace | Standard Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/37
Other Adverse Events (participants affected / at risk) | 0/62 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT05037578/Prot_SAP_ICF_000.pdf